CLINICAL TRIAL: NCT02243605
Title: A Phase 2 Study of XL184 (Cabozantinib) in Treating Patients With Relapsed Osteosarcomas and Ewing Sarcomas
Brief Title: Cabozantinib S-malate in Treating Patients With Relapsed Osteosarcoma or Ewing Sarcoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2014-01927; NCI-2014-01927 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CABONE; 9620 (Other: Institut Bergonie Cancer Center); 9620 (Other: CTEP)
Record Dates: First submitted 2014-09-16; First posted 2014-09-18 (Estimated); Results first posted 2020-09-04 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-06

CONDITIONS: Metastatic Ewing Sarcoma; Metastatic Osteosarcoma; Recurrent Ewing Sarcoma; Recurrent Osteosarcoma; Stage III Osteosarcoma AJCC v7; Stage IV Osteosarcoma AJCC v7; Stage IVA Osteosarcoma AJCC v7; Stage IVB Osteosarcoma AJCC v7; Unresectable Ewing Sarcoma; Unresectable Osteosarcoma
MeSH Terms: conditions — Sarcoma, Ewing; Osteosarcoma | interventions — cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (cabozantinib s-malate) (Experimental): Patients receive cabozantinib s-malate PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cabozantinib S-malate; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Cabozantinib S-malate — Given PO
  Other Names: BMS-907351; Cabometyx; Cometriq; XL 184; XL-184; XL184
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial studies how well cabozantinib s-malate works in treating patients with osteosarcoma or Ewing sarcoma that has grown or returned (come back) after a period of improvement. Cabozantinib s-malate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and may also prevent the growth of new blood vessels that tumors need to grow.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the antitumor activity of cabozantinib s-malate (cabozantinib) for Ewing sarcomas, in terms of 6-month objectives response as per the Response Evaluation Criteria in Solid Tumors, Revised (RECIST version [v]1.1).

II. To evaluate the antitumor activity of cabozantinib for osteosarcoma, in terms of 6-month objective response (complete response, partial response) and 6-month non-progression (complete response, partial response and stable disease), as per RECIST v1.1.

SECONDARY OBJECTIVES:

I. 6-month objective response. (Ewing sarcoma only) II. Best overall response (as per the revised RECIST v1.1). (Ewing sarcoma and osteosarcoma) III. 1- and 2-year progression-free survival. (Ewing sarcoma and osteosarcoma) IV. 1- and 2-year overall survival. (Ewing sarcoma and osteosarcoma) V. Cabozantinib safety. (Ewing sarcoma and osteosarcoma) VI. To assess the ability of metabolic tumor response as measured by fludeoxyglucose (FDG)-positron emission tomography (PET) at the end of one cycle of treatment to predict progression-free survival (PFS). (Ewing sarcoma and osteosarcoma) VII. Translational research: to determine and compare tumor expression of MET, phosphorylated (phosphor)-MET and circulating levels of HGF, soluble MET (sMET), VEGF-A, and soluble VEGF receptor 2 (VEGFR2) (sVEGFR2) prior to and following administration of cabozantinib. (Ewing sarcoma and osteosarcoma)

OUTLINE:

Patients receive cabozantinib s-malate orally (PO) once daily (QD) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Young patient age between 12 - 15 could be included in only 6 centers (Bordeaux, Lyon, Villejuif, Lille, Marseille and Paris)
* Patients must have histologically confirmed diagnosis of osteosarcoma or Ewing sarcoma by central review, except if the diagnosis was already confirmed by the RRePS (Reseau de Reference en Pathologie des Sarcomes et des Tissus Mous et des Visceres) network
* Relapsed disease after standard chemotherapy
* Patients must have measurable disease (lesion in previously irradiated field could be considered as measurable if progressive at inclusion) defined as per RECIST v1.1 with at least one lesion that can be measured in at least one dimension (longest diameter to be recorded) as >= 10 mm with spiral computed tomography (CT) scan
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1
* Life expectancy of greater than 3 months
* Absolute neutrophil count >= 1,500/mcL
* Lymphocyte count > 1,000/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3.0 x institutional upper limit of normal
* Creatinine =< 1.5 x ULN OR creatinine clearance >= 50 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal (Cockcroft formula)
* Hemoglobin >= 9 g/dL
* Serum albumin >= 2.8 g/dL
* Lipase < 2.0 x ULN and no radiologic or clinical evidence of pancreatitis
* Urine protein/creatinine ratio (UPCR) =< 1
* Serum phosphorus >= lower limit of normal (LLN)
* Serum calcium >= LLN
* Serum magnesium >= LLN
* Serum potassium >= LLN
* Female subjects of childbearing potential must not be pregnant at screening; females of childbearing potential are defined as premenopausal females capable of becoming pregnant (ie, females who have had any evidence of menses in the past 12 months, with the exception of those who had prior hysterectomy); however, women who have been amenorrheic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, antiestrogens, low body weight, ovarian suppression or other reasons
* The effects of Cabozantinib on the developing human fetus are unknown; for this reason and because tyrosine kinase inhibitors agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (see below) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of cabozantinib administration

  * Sexually active subjects (men and women) must agree to use medically accepted barrier methods of contraception (e.g., male or female condom) during the course of the study and for 4 months after the last dose of study drug(s), even if oral contraceptives are also used; all subjects of reproductive potential must agree to use both a barrier method and a second method of birth control during the course of the study and for 4 months after the last dose of study drug(s)
* Metastatic or unresectable locally advanced
* Documented disease progression (as per RECIST v1.1) before study entry; for patients with osteosarcoma, this progression will be confirmed by central review on the basis of two CT scan or magnetic resonance imaging (MRI) obtained at less than 6 months in the period of 12 months prior to inclusion
* Ability to understand and the willingness to sign a written informed consent document
* In accordance with French Regulatory Authorities: Patients with French Social Security in compliance with the French law relating to biomedical research (Huriet Law 88-1138 and related decrees)

Exclusion Criteria:

* The subject has received cytotoxic chemotherapy (including investigational cytotoxic chemotherapy) or biologic agents (e.g., cytokines or antibodies) within 3 weeks, or nitrosoureas/mitomycin C within 6 weeks before the first dose of study treatment
* Prior treatment with cabozantinib
* Radiation therapy for bone metastasis within 2 weeks, any other external radiation therapy within 4 weeks before the first dose of study treatment; systemic treatment with radionuclides within 6 weeks before the first dose of study treatment; subjects with clinically relevant ongoing complications from prior radiation therapy are not eligible
* Receipt of any type of small molecule kinase inhibitor (including investigational kinase inhibitor) within 14 days before the first dose of study treatment; note: subjects with prostate cancer currently receiving luteinizing hormone-releasing hormone (LHRH) or gonadotropin-releasing hormone (GnRH) agonists may be maintained on these agents
* The subject has received any other type of investigational agent within 28 days before the first dose of study treatment
* The subject has not recovered to baseline or Common Terminology Criteria for Adverse Events (CTCAE) =< grade 1 from toxicity due to all prior therapies except alopecia and other non-clinically significant adverse events (AEs)
* The subject has a primary brain tumor
* Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 2 weeks before the first dose of study treatment; eligible subjects must be neurologically asymptomatic and without corticosteroid treatment at the time of the start of study treatment
* The subject has prothrombin time (PT)/international normalized ratio (INR) or partial thromboplastin time (PTT) test >= 1.3 x the laboratory ULN within 7 days before the first dose of study treatment
* The subject requires concomitant treatment, in therapeutic doses, with anticoagulants such as warfarin or warfarin-related agents, heparin, thrombin or factor Xa inhibitors, or antiplatelet agents (e.g., clopidogrel); low dose aspirin (=< 81 mg/day), low-dose warfarin (=< 1 mg/day), and prophylactic low molecular weight heparin (LMWH) are permitted
* The subject requires chronic concomitant treatment of strong cytochrome P450 family 3, subfamily A, polypeptide 4 (CYP3A4) inducers (e.g., dexamethasone, phenytoin, carbamazepine, rifampin, rifabutin, rifapentine, phenobarbital, and St. John's wort)

  * it is important to regularly consult a frequently-updated list; medical reference texts such as the Physicians' Desk Reference may also provide this information; as part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* The subject has experienced any of the following:

  * Clinically-significant gastrointestinal bleeding within 6 months before the first dose of study treatment
  * Hemoptysis of >= 0.5 teaspoon (2.5 mL) of red blood within 3 months before the first dose of study treatment
  * Any other signs indicative of pulmonary hemorrhage within 3 months before the first dose of study treatment
* The subject has radiographic evidence of cavitating pulmonary lesion(s)
* The subject has tumor in contact with, invading or encasing any major blood vessels
* The subject has evidence of tumor invading the gastrointestinal (GI) tract (esophagus, stomach, small or large bowel, rectum or anus), or any evidence of endotracheal or endobronchial tumor within 28 days before the first dose of cabozantinib
* The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

  * Cardiovascular disorders including:

    * Congestive heart failure (CHF): New York Heart Association (NYHA) class III (moderate) or class IV (severe) at the time of screening
    * Concurrent uncontrolled hypertension defined as sustained blood pressure (BP) > 150 mm Hg systolic, or > 90 mm Hg diastolic despite optimal antihypertensive treatment within 7 days of the first dose of study treatment
    * Any history of congenital long QT syndrome
    * Any of the following within 6 months before the first dose of study treatment:

      * Unstable angina pectoris
      * Clinically-significant cardiac arrhythmias
      * Stroke (including transient ischemic attack [TIA], or other ischemic event)
      * Myocardial infarction
      * Thromboembolic event requiring therapeutic anticoagulation (note: subjects with a venous filter [e.g. vena cava filter] are not eligible for this study)
  * Gastrointestinal disorders particularly those associated with a high risk of perforation or fistula formation including:

    * Any of the following within 28 days before the first dose of study treatment

      * Intra-abdominal tumor/metastases invading GI mucosa
      * Any evidence of active peptic ulcer disease, patients must be completely recovered
      * Any evidence of inflammatory bowel disease (including ulcerative colitis and Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, patients must be completely recovered from these conditions
      * Malabsorption syndrome
    * Any of the following within 6 months before the first dose of study treatment:

      * Abdominal fistula
      * Gastrointestinal perforation
      * Bowel obstruction or gastric outlet obstruction
      * Intra-abdominal abscess; note: complete resolution of an intra-abdominal abscess must be confirmed prior to initiating treatment with cabozantinib even if the abscess occurred more than 6 months before the first dose of study treatment
  * Other disorders associated with a high risk of fistula formation including percutaneous endoscopic gastrostomy (PEG) tube placement within 3 months before the first dose of study therapy
  * Other clinically significant disorders such as:

    * Active infection requiring systemic treatment within 28 days before the first dose of study treatment
    * Serious non-healing wound/ulcer/bone fracture within 28 days before the first dose of study treatment
    * History of organ transplant
    * Concurrent uncompensated hypothyroidism or thyroid dysfunction within 7 days before the first dose of study treatment
    * History of major surgery as follows:

      * Major surgery within 12 weeks before the first dose of study treatment; complete wound healing from major surgery must have occurred 1 month before the first dose of study treatment
      * Minor surgery (including uncomplicated tooth extractions) within 28 days before the first dose of study treatment with complete wound healing at least 10 days before the first dose of study treatment; subjects with clinically relevant ongoing complications from prior surgery are not eligible
* The subject is unable to swallow tablets
* The subject has a corrected QT interval calculated by the Fridericia formula (QTcF) > 500 ms within 28 days before treatment; note: if initial QTcF is found to be > 500 ms, two additional electrocardiograms (EKGs) separated by at least 3 minutes should be performed; if the average of these three consecutive results for QTcF is =< 500 ms, the subject meets eligibility in this regard
* The subject is unable or unwilling to abide by the study protocol or cooperate fully with the investigator or designee
* The subject has had evidence within 2 years of the start of study treatment of another malignancy which required systemic treatment
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to cabozantinib
* Pregnant women are excluded from this study because cabozantinib is a tyrosine kinase inhibitor with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with cabozantinib, breastfeeding should be discontinued if the mother is treated with cabozantinib; these potential risks may also apply to other agents used in this study
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with cabozantinib; in addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated
* Participation to a study involving a medical or therapeutic intervention in the last 30 days
* Prior participation in this study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2014-12-19 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2026-07-11 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Italiano, Principal Investigator — Institut Bergonie Cancer Center
Locations (11):
- France (11):
  - Institut Bergonie Cancer Center, Bordeaux
  - Centre Georges-Francois Leclerc, Dijon
  - Centre Oscar Lambert, Lille
  - Centre Leon Berard, Lyon
  - Hopital De La Timone, Marseille
  - Centre Antoine Lacassagne, Nice
  - Institut Curie Paris, Paris
  - Institut de Cancerologie de l'Ouest-Rene Gauducheau, Saint-Herblain
  - CHRU Strasbourg - Hospital Civil, Strasbourg
  - Center Claudius Regaud, Toulouse
  - Gustave Roussy, Villejuif

REFERENCES:
- [Derived] Italiano A, Mir O, Mathoulin-Pelissier S, Penel N, Piperno-Neumann S, Bompas E, Chevreau C, Duffaud F, Entz-Werle N, Saada E, Ray-Coquard I, Lervat C, Gaspar N, Marec-Berard P, Pacquement H, Wright J, Toulmonde M, Bessede A, Crombe A, Kind M, Bellera C, Blay JY. Cabozantinib in patients with advanced Ewing sarcoma or osteosarcoma (CABONE): a multicentre, single-arm, phase 2 trial. Lancet Oncol. 2020 Mar;21(3):446-455. doi: 10.1016/S1470-2045(19)30825-3. Epub 2020 Feb 17. PMID 32078813
- [Derived] Hattinger CM, Patrizio MP, Magagnoli F, Luppi S, Serra M. An update on emerging drugs in osteosarcoma: towards tailored therapies? Expert Opin Emerg Drugs. 2019 Sep;24(3):153-171. doi: 10.1080/14728214.2019.1654455. Epub 2019 Aug 14. PMID 31401903

RESULTS

PARTICIPANT FLOW:
Groups:
- Ewing Sarcoma: Patients receive cabozantinib s-malate PO QD on days 1-28. 60 mg for patients ≥ 16 years and 40mg/m² for patients ≥ 12 years and <16 years. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Single-arm phase II clinical trial based on a two-stage optimal Simon's design with 41 evaluable patients (first stage: 21 patients) used to distinguish a favorable true objective response rate within 6 months of treatment onset of 20% from a null rate of 5% (90% power and 5% type I error).
  Stage 1(21 evaluable patients): if <=1 objective response within 6 months of treatment onset, the study was stopped early. Otherwise, the second group of 20 participants was recruited.
  Stage 2 (41 evaluable patients): if >= 5 objective response within 6 months of treatment onset, Cabozantinib was considered promising.
- Osteosarcoma: Patients receive cabozantinib s-malate PO QD on days 1-28. 60 mg for patients ≥ 16 years and 40mg/m² for patients ≥ 12 years and <16 years. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Single-arm phase II trial based on 2-stage dual endpoint design with 41 evaluable patients (first stage: 21 patients) used to distinguish :
  * a favorable true 6-month non-progression rate of 50% from a null rate of 25% (92% power).
  * a favorable true objective response rate within 6 months of treatment onset of 20% from a null rate of 5% (90% power).
  Stage 1(21 evaluable patients): if <=1 objective response within 6 months of treatment onset or <=6 6-month non-progression, the study was stopped early. Otherwise, the second group of 20 participants was recruited.
  Stage 2 (41 evaluable patients): if >= 5 objective response within 6 months of treatment onset or >=16 6-month non-progression, Cabozantinib was considered promising.
Period: Stage 1 - Interim Analysis Population
Arm/Group | Ewing Sarcoma | Osteosarcoma
Started | 23 | 22
Completed (Eligible and who received at least one complete cycle or two incomplete cycles of treatment.) | 21 | 21
Not Completed | 2 | 1
Not completed — Protocol Violation | 1 | 1
Not completed — Adverse Event | 1 | 0
Period: Stage 2 - Final Analysis Population
Arm/Group | Ewing Sarcoma | Osteosarcoma
Started | 45 | 45
Completed (Eligible and who received at least one complete cycle or two incomplete cycles of treatment.) | 39 | 42
Not Completed | 6 | 3
Not completed — Protocol Violation | 5 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Progression | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ewing Sarcoma | Osteosarcoma | Total
Number analyzed (Participants) | 45 | 45 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 7 | 13
  Between 18 and 65 years | 38 | 31 | 69
  >=65 years | 1 | 7 | 8
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 33 [24 to 45] | 34 [20 to 53] | 34 [21 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 18 | 32
  Male | 31 | 27 | 58
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 45 | 45 | 90

OUTCOME MEASURES:

1. Primary Outcome: Non-progression at 6 Months - Osteosarcoma
Description: Non-progression defined as complete response (CR), partial response (PR), or stable disease (SD) as per the Response Evaluation Criteria In Solid Tumors Criteria, revised RECIST v1.1.
  As per revised RECIST v1.1, progression is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study, or a measurable increase in a non-target lesion, or the appearance of one or more new lesions.
Time Frame: At 6 months
Population: All patients eligible and who received at least one complete or two incomplete treatment cycles.
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Osteosarcoma
Number analyzed (Participants) | 42
percentage | 33.3 [19.6 to 49.6]

2. Primary Outcome: Objective Response Within 6 Months of Treatment Onset - Osteosarcoma
Description: Objective response defined as complete response (CR) or partial response (PR) as per the Response Evaluation Criteria In Solid Tumors Criteria, revised RECIST v1.1.
  As per revised RECIST v1.1, CR is defined as disappearance of all target and non-target lesions and normalization of tumour marker level of non-target lesions. All lymph nodes must be non-pathological in size (<10 mm short axis).
  As per revised RECIST v1.1, PR is defined as a at least 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters, and non-PD/not all evaluated non-target lesions, or, CR of target lesions and non-CR/non-PD/not evaluated non-target lesions.
  As per revised RECIST v1.1, progression is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study, or a measurable increase in a non-target lesion, or the appearance of one or more new lesions.
Time Frame: Within 6 months of treatment onset
Population: All patients eligible and who received at least one complete or two incomplete treatment cycles.
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Osteosarcoma
Number analyzed (Participants) | 42
percentage | 11.9 [4.0 to 25.6]

3. Primary Outcome: Objective Response Within 6 Months of Treatment Onset - Ewing Sarcoma
Description: as for outcome 2
Time Frame: Within 6 months of treatment onset
Population: All patients eligible and who received at least one complete or two incomplete treatment cycles.
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Ewing Sarcoma
Number analyzed (Participants) | 39
percentage | 25.6 [13.0 to 42.1]

4. Secondary Outcome: Best Overall Response
Description: Best objective response rate, defined as the rate of CR or PR confirmed ≥ 4 weeks after initial documentation, as determined by investigator review of tumor assessments using RECIST v1.1. Complete or partial responses may be claimed only if the criteria for each are met at a subsequent time point as specified in the protocol (generally 4 weeks later). The BOR is the best response recorded from the start of the study treatment until the end of treatment
  * Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm
  * Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters
  * Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions and also demonstrate an absolute increase of at least 5 mm
  * Stable Disease (SD): Neither sufficient shrinkage to qualify for PR
Time Frame: From the start of the treatment until disease progression/recurrence. assessed up to 2 years.
Population: All patients eligible and who received at least one complete or two incomplete treatment cycles.
Measure: Count of Participants; unit: Participants
Arm/Group | Ewing Sarcoma | Osteosarcoma
Number analyzed (Participants) | 39 | 42
Participants
  Partial response | 5 | 3
  Stable disease | 19 | 21
  Progressive disease | 12 | 15
  Not evaluable | 3 | 3

5. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the duration of time from start of treatment to time of progression (clinical and/or radiological) or death, whichever occurs first. Radiological progression is assessed by local review of tumor assessments using RECIST v1.1 criteria : at least a 20% increase in the sum of the diameters of target lesions and also demonstrate an absolute increase of at least 5 mm.
Time Frame: Time from start of treatment to time of progression or death, whichever occurs first, assessed up to 2 years
Population: All patients eligible and who received at least one complete or two incomplete treatment cycles.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ewing Sarcoma | Osteosarcoma
Number analyzed (Participants) | 39 | 42
months | 4.4 [3.7 to 5.6] | 5.9 [4.7 to 7.4]

6. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the duration of time from start of treatment to the time of death.
Time Frame: Time from start of treatment to the time of death, assessed up to 2 years
Population: All patients eligible and who received at least one complete or two incomplete treatment cycles.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ewing Sarcoma | Osteosarcoma
Number analyzed (Participants) | 39 | 42
months | 12.5 [8.5 to 20.7] | 10.4 [7.4 to 12.5]

7. Secondary Outcome: Non-progression at 6 Months - Ewing Sarcoma
Description: as for outcome 1
Time Frame: At 6 months
Population: All patients eligible and who received at least one complete or two incomplete treatment cycles.
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Ewing Sarcoma
Number analyzed (Participants) | 39
percentage | 25.6 [13.0 to 42.1]

8. Secondary Outcome: Incidence of Adverse Events
Description: Number of patients who had at least one adverse event related to the treatment. Adverse events were assessed using CTCAE (5.0).
Time Frame: Safety profile was continuously followed during treatment and up to 30 days after the last Cabozantinib dose or until the start of a new antitumor therapy, whichever occurs first.
Population: Adverse event are reported for all treated patients who received at least one administration of treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Osteosarcoma; Ewing Sarcoma: Patients receive cabozantinib s-malate PO QD on days 1-28. 60 mg for patients ≥ 16 years and 40mg/m² for patients ≥ 12 years and <16 years. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | Osteosarcoma | Ewing Sarcoma
Number analyzed (Participants) | 45 | 45
Participants | 45 | 45

ADVERSE EVENTS:
Time Frame: Safety profile was continuously followed during treatment and up to 30 days after the last Cabozantinib dose or until the start of a new antitumor therapy, whichever occurs first.
Description: Adverse event are reported for all treated patients who received at least one administration of treatment.
  All adverse events (related and unrelated to treatment) are reported. All serious adverse events (related and unrelated to treatment) are reported.
Arm/Group | Osteosarcoma | Ewing Sarcoma
All-Cause Mortality (participants affected / at risk) | 42/45 | 37/45
Serious Adverse Events (participants affected / at risk) | 30/45 | 31/45
Other Adverse Events (participants affected / at risk) | 45/45 | 45/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Osteosarcoma (N=45) | Ewing Sarcoma (N=45)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 2 (2) | 1 (1)
Hypocinetic cardiopathy (Cardiac disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peritoneal effusion (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death NOS (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 1 (1)
Worsening of general status (General disorders) | 2 (2) | 3 (3)
Thoracic pain (General disorders) | 0 (0) | 1 (1)
Disease progression (General disorders) | 2 (2) | 4 (4)
Icteric cholestasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anorectal infection (Infections and infestations) | 0 (0) | 1 (1)
Bronchial infection (Infections and infestations) | 1 (1) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0)
Localized infection (Infections and infestations) | 0 (0) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
GGT increased (Investigations) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 1 (1) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Pancytopenia (Investigations) | 0 (0) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetes (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (3)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast microcalcification presence (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Medullary compression (Nervous system disorders) | 1 (1) | 1 (1)
Deficit of lower limbs (Nervous system disorders) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 2 (2)
Relapse of psychiatric disorders (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 9 (11) | 10 (14)
Pneumopathy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumomediatinum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Skin ulceration (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Thromboembolic event (Vascular disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Osteosarcoma (N=45) | Ewing Sarcoma (N=45)
Anemia (Blood and lymphatic system disorders) | 5 (7) | 6 (7)
Sinus tachycardia (Cardiac disorders) | 3 (3) | 4 (4)
Hypothyroidism (Endocrine disorders) | 23 (25) | 21 (23)
Blurred vision (Eye disorders) | 1 (1) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 8 (10) | 12 (12)
Constipation (Gastrointestinal disorders) | 14 (21) | 14 (17)
Diarrhea (Gastrointestinal disorders) | 31 (47) | 33 (51)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 7 (8)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 4 (4)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 (3) | 7 (8)
Gastrointestinal disorders - Other, specify : gastroenteritis (Gastrointestinal disorders) | 3 (3) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 3 (3) | 5 (6)
Hemorrhoids (Gastrointestinal disorders) | 2 (2) | 3 (3)
Mucositis oral (Gastrointestinal disorders) | 26 (32) | 24 (31)
Nausea (Gastrointestinal disorders) | 19 (22) | 15 (19)
Periodontal disease (Gastrointestinal disorders) | 3 (5) | 4 (6)
Toothache (Gastrointestinal disorders) | 4 (4) | 2 (2)
Vomiting (Gastrointestinal disorders) | 7 (9) | 10 (12)
Fatigue (General disorders) | 33 (41) | 32 (36)
Fever (General disorders) | 8 (11) | 6 (8)
Non-cardiac chest pain (General disorders) | 7 (11) | 4 (4)
Pain (General disorders) | 6 (7) | 5 (5)
Bronchial infection (Infections and infestations) | 4 (7) | 3 (4)
Pharyngitis (Infections and infestations) | 2 (2) | 4 (4)
Rhinitis infective (Infections and infestations) | 4 (4) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 4 (5)
Urinary tract infection (Infections and infestations) | 3 (3) | 3 (5)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Alanine aminotransferase increased (Investigations) | 21 (25) | 22 (27)
Alkaline phosphatase increased (Investigations) | 6 (6) | 7 (9)
Aspartate aminotransferase increased (Investigations) | 22 (28) | 22 (27)
Blood bilirubin increased (Investigations) | 3 (3) | 3 (3)
Blood lactate dehydrogenase increased (Investigations) | 7 (10) | 7 (8)
CPK increased (Investigations) | 1 (1) | 4 (7)
Electrocardiogram QT corrected interval prolonged (Investigations) | 4 (4) | 0 (0)
GGT increased (Investigations) | 2 (2) | 4 (4)
Lipase increased (Investigations) | 6 (18) | 4 (5)
Lymphocyte count decreased (Investigations) | 2 (5) | 4 (7)
Neutrophil count decreased (Investigations) | 7 (10) | 9 (11)
Platelet count decreased (Investigations) | 14 (16) | 16 (19)
Serum amylase increased (Investigations) | 4 (4) | 2 (2)
Thyroid stimulating hormone increased (Investigations) | 6 (6) | 4 (4)
Weight loss (Investigations) | 14 (15) | 14 (14)
White blood cell decreased (Investigations) | 3 (6) | 5 (7)
Anorexia (Metabolism and nutrition disorders) | 23 (27) | 11 (13)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 6 (9) | 4 (5)
Hypokalemia (Metabolism and nutrition disorders) | 8 (14) | 6 (6)
Hypomagnesemia (Metabolism and nutrition disorders) | 11 (18) | 7 (9)
Hypophosphatemia (Metabolism and nutrition disorders) | 10 (12) | 14 (23)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (8) | 11 (14)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (8) | 7 (9)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (8) | 6 (7)
Dysesthesia (Nervous system disorders) | 3 (3) | 2 (2)
Dysgeusia (Nervous system disorders) | 9 (10) | 15 (15)
Headache (Nervous system disorders) | 7 (10) | 10 (12)
Anxiety (Psychiatric disorders) | 5 (5) | 2 (2)
Depression (Psychiatric disorders) | 5 (5) | 2 (2)
Insomnia (Psychiatric disorders) | 6 (6) | 3 (3)
Proteinuria (Renal and urinary disorders) | 7 (9) | 4 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (14) | 10 (13)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 5 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 4 (5)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 5 (5)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (6) | 6 (6)
Dry skin (Skin and subcutaneous tissue disorders) | 13 (15) | 16 (17)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 3 (4) | 3 (3)
Hair color changes (Skin and subcutaneous tissue disorders) | 18 (18) | 16 (16)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 12 (13) | 17 (21)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify: Erythema (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1) — Osteosarcoma : 1 ERYTHEMA, 1 LEFT KNEE SCAR ERYTHEMA, 1 SCALP ERYTHEMA, 1 SOLAR ERYTHEMA Ewing sarcoma : 1 STUMP ERYTHEMA
Skin and subcutaneous tissue disorders - Other, specify: Ungual hemorrhage (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) — Osteosarcoma : 1 NAIL HEMORRHAGE, 1 SUBUNGUAL HEMORRHAGE, 1 UNGUAL HEMORRHAGE
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 6 (6) | 5 (5)
Skin ulceration (Skin and subcutaneous tissue disorders) | 4 (6) | 2 (2)
Hypertension (Vascular disorders) | 7 (9) | 3 (3)
Thromboembolic event (Vascular disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-04): https://cdn.clinicaltrials.gov/large-docs/05/NCT02243605/Prot_SAP_000.pdf